CLINICAL TRIAL: NCT07256210
Title: Phase I/II Clinical Trial of mbIL21 ex Vivo-expanded Donor-derived NK-cell Infusions With Hematopoietic Stem Cell Transplantation for Disease Relapse Prophylaxis in Pediatric and Young Adult Patients With Chemorefractory or Minimal Residual Disease Positive Acute Leukemia
Brief Title: Feasibility and Safety of Donor-derived NK-cell Infusions for Leukemia Relapse Prophylaxis After Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NDGOI-11-2024
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic T-cell Leukemia; Mixed Phenotype Acute Leukemia
Keywords: Natural killer cell therapy; Hematopoietic stem cell transplantation; Leukemia, Acute; Refractory Leukemias; Pre-transplantation MRD-positivity
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological: Donor-derived Natural Killer Cell Infusions (Experimental)
  Interventions: Biological: Donor-derived Natural Killer Cell

INTERVENTIONS:
Biological: Donor-derived Natural Killer Cell — These are total doses for two infusions. The first NK-cell infusion on day -12 comprises 2/3 of total NK-cell dose and the second NK-cell infusion approximately on day +5 consists of 1/3 of total NK-cell dose.

SUMMARY:
This pilot clinical trial aims to evaluate the feasibility, adverse reactions and maximum tolerated dose of mbIL21 ex vivo-expanded donor-derived NK-cell infusions before and after haploidentical or matched-related hematopoietic stem cell transplantation in a cohort of pediatric and young adult patients with chemorefractory or minimal residual disease (MRD) positive acute leukemia.

DETAILED DESCRIPTION:
Rationale. In the context of treating children and young adults with high-risk or chemorefractory acute leukemia allogeneic hematopoietic stem cell transplantation (allo-HSCT) plays a crucial role. It is well known, that residual tumor cell volume at the time of allo-HSCT has a significant impact on its outcomes. The antileukemic effect of allo-HSCT in some hematologic malignancies is predominantly mediated by graft-versus-leukemia effect, which is an immune-mediated reaction of engrafted donor hematopoiesis against the recipient's tumor cells. The graft-versus-leukemia effect is generally ascribed to NK-cells conserved within the graft or arising from it early after transplantation.

Primary objective: to evaluate feasibility, safety and to identify the maximum tolerated dose (MTD) of mbIL21 ex vivo-expanded donor-derived NK-cell cells to be infused to children and young adults aged 1 to 25 years with chemorefractory or pre-transplant MRD-positive acute leukemia undergoing allo-HSCT.

Secondary objectives:

1. To assess the short-term disease response to NK cell infusions as an adjunct to allo-HSCT.
2. To assess the impact of NK cell infusions on reconstitution of main lymphocyte subpopulations in allo-HSCT recipients.
3. To assess the impact of NK cell infusions on main allo-HSCT outcomes. Outline. This is a phase I, 3+3 dose-escalation study of NK-cells followed by a phase II study. Conditioning regimen will be split into two parts. Two donor NK-cell infusions will be carried out: after the first part of conditioning and early after transplant.

FIRST PART OF CONDITIONING: Patients receive fludarabine 40 mg/m2/day IV over 1 hour on days -14 and -13, thiotepa 10 mg/kg/course IV over 1 hour on days -14 and -13 and cyclophosphamide 500 mg/m2 IV over 1 hour on day -14.

SECOND PART OF CONDITIONING: Patients receive fludarabine 40 mg/m2/day IV over 1 hour on days -4 and -3, treosulfan 42 g/m2/course IV over 2 hours on days -4, -3, -2 or busulfan 12 mg/kg/course PO on days -4, -3, -2 or total body irradiation (TBI) 12 Gy/course on days -4, -3, -2.

TRANSPLANT: Patients undergo allogeneic G-CSF mobilized CD3-depleted peripheral blood stem cell transplantation on day 0.

PHARMACOLOGIC GVHD PROPHYLAXIS: Patients receive tocilizumab 8 mg/kg on day -1 and abatacept 10 mg/kg/day IV over 1 hour on days -1, +7, +14 and +28 (the last one - only in case of haploidentical donor).

DONOR NK-CELL INFUSIONS: Each patient is planned to receive two mbIL21 ex vivo-expanded donor-derived NK-cell infusions. Escalating doses of NK-cells (CD3-CD56+) to be infused in the Phase I study as follows:

* Level 1: 10х106/kg
* Level 2: 20х106/kg
* Level 3: 30х106/kg In case of level 1 dose is not tolerated, an additional dose level (Level 0 - 5х106/kg) can be added. In the absence of unacceptable toxicity level 1 dose further can be used.

These are total doses for two infusions. The first NK-cell infusion on day -12 comprises 2/3 of total NK-cell dose and the second NK-cell infusion approximately on day +5 consists of 1/3 of total NK-cell dose.

To be able to receive NK-cell infusion patient must fulfil the following clinical criteria:

1. Off corticosteroids more than 0,5 mg/kg/day prednisone or equivalent within prior 72 hours period;
2. No uncontrolled infection within 24 hours;
3. No grade 3 or greater nonhematologic adverse reactions (only for the second NK-cell infusion);
4. Not requiring ventilator support or more than 5 L/min of supplemental oxygen. DONOR SELECTION CRITERIA: In case of detection of two or more suitable donors, besides standart donor selection criteria (CMV serology, sex, blood group etc.) the choice will be made in favor of the presence of KIR-ligand mismatch.

DURATION OF THERAPY: 21 day (14 days before HSCT and up to 7 days after HSCT). Follow up during 2 years after HSCT.

CRITERIA FOR PREMATURE STOPPING OF THE STUDY: DLT in 2 patients of expanded cohort with a minimum (Level 0) dose level. DLT is defined as associated with the intervention immune-related adverse event (cytokine release syndrome or immune effector cell-associated neurotoxicity syndrome) grade 3 or higher according to ASTCT criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (age from 14 to 25 years) and/or patient's legal representative (age from 0 to 18 years) should provide written informed consent.
2. Patients with one of the following disease:

   * Acute myeloid leukemia: a. primary refractory disease (absence of complete remission (CR) after two induction regimens), b. refractory relapse (absence of CR after one salvage regimen), c. MRD-persistence before conditioning (presence of residual leukemic population more than 0,01% of bone marrow nucleated cells by flow cytometry);
   * Acute T-lymphoblastic leukemia: a. primary refractory disease (absence of complete remission (CR) after two induction regimens), b. refractory relapse (absence of CR after one salvage regimen), c. MRD-persistence before conditioning (presence of residual leukemic population more than 0,1% of bone marrow nucleated cells by flow cytometry);
   * Acute mixed phenotype leukemia: a. primary refractory disease (absence of complete remission (CR) after two induction regimens), b. refractory relapse (absence of CR after one salvage regimen), c. MRD-persistence before conditioning (presence of residual leukemic population more than 0,01% of bone marrow nucleated cells by flow cytometry).
3. Patient is indicated to receive allo-HSCT according to actual clinical practice.
4. Haploidentical or matched related donor was chosen and is available for allo-HSCT (and NK-cell therapy).
5. Patient's clinical status: Lansky/Karnowski index ≥50%.
6. Kidney function: clearance of endogenous creatinine or glomerular filtration rate according to Schwarz equation ≥50 ml/min/1,73 m2.
7. Liver function: total bilirubin ≤3 ULN except for Gilbert's disease, ALT/AST ≤3 ULN.
8. Heart function: left ventricular ejection fraction ≥40%.
9. Lung function: lung capacity ≥50%, for children who cannot carry out of respiratory function - oxygen saturation during pulse oximetry ≥92% (without supplemental oxygen).
10. Life expectancy ≥8 weeks.
11. Patients who agree to long-term follow up for up to 2 years.

Exclusion Criteria:

1. Inability to provide or withdrawal of written informed consent.
2. Cellular therapy including allo-HSCT within prior 4 months period, absence of active signs of GVHD, sinusoidal obstruction syndrome, cytokine release syndrome, immune effector cell-associated neurotoxicity syndrome.
3. Active hepatitis B, C or HIV infection.
4. Pregnant or lactating women.
5. Uncontrolled infection; principal investigator is the final arbiter of this criterion.
6. Clinical signs of grade ≥3 CNS disorders (seizure disorder, paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injuries, dementia, organic brain syndrome, psychosis, coordination or movement disorder).
7. Mental illness of the patient or caregivers, making it impossible to realize the essence of the study and compromising compliance with medical appointments and sanitary and hygienic regime.

Ages: 1 Month to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who received the planned dose of NK cells without adverse reactions grade ≥3 according to CTCAE v5.0 | 180 days from the last administration of donor NK cells

SECONDARY OUTCOMES:
Rate of morphologic bone marrow leukemia-free state | on day -4 before HSCT, and +30 days after HSCT
  Rate of morphologic bone marrow leukemia-free state on day -4, morphologic complete remission on day +30 (only for patients with chemorefractory acute leukemia).
Rate of MRD-negativity | on days -4 before HSCT and +30 days after HSCT
Cumulative incidence of developing acute graft-versus-host disease | 180 days from the last administration of donor NK cells
Cumulative incidence of relapse | 2 years after allo-HSCT
Cumulative incidence of transplantation-related mortality | 100 days and 2 years after allo-HSCT
Probability of engraftment | 30 days after allo-HSCT
Overall survival | 2 years after allo-HSCT

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev Federal Research and Clinical Centre of Paediatric Haematology, Oncology and Immunology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No